CLINICAL TRIAL: NCT00768443
Title: Epidemiological Study to Assess the Symptom Patterns and Management Strategies in Patients Consulting With Persistent GERD Symptoms in Primary Care
Brief Title: Symptoms and Management Strategies in Gastroesophageal Reflux Disease (GERD)
Acronym: PHENIX
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-GHR-NEX-2008/1
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; PPI
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This a non-interventional multi-centre study to evaluate the symptom load and management strategies in PPI-treated GERD patients with persistent GERD symptoms..

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Subjects with a diagnosis of GERD and with predominant typical GERD symptoms: heartburn/regurgitation
* Subjects who fail to obtain satisfactory symptomatic response after their first full course (4-8 weeks) of standard dose PPI (once a day)

Exclusion Criteria:

* Inability to read and/or understand Patient Reported Outcomes questionnaires
* Subjects where the only reason for the visit is renewing the prescription
* A history of an incomplete response to PPI treatment prior to current course of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PPI-treated patients consulting with persistent GERD symptoms in Primary Care. The patients must have a diagnosis of GERD with predominant typical GERD symptoms and fail to obtain satisfactory symptomatic response after the first full course of standard dose PPI. The patients must have been on continuous PPI treatment with unchanged doses according to local labelling during the last 4-8 weeks prior to the enrolment visit.
Sampling Method: Non-Probability Sample
Enrollment: 2674 (Actual)
Dates: Start 2008-09; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To assess the symptom load and impact on daily life in PPI-treated GERD patients with persistent GERD symptoms | Once, at first visit

SECONDARY OUTCOMES:
To describe the frequency and severity of extra-oesophageal and/or atypical GERD symptoms and to assess the concordance between patient-reported and physician-reported symptom load | Once, at first visit
To describe current and previous treatment strategies and to describe the diagnostic and therapeutic approaches during the study visit | Once, at first visit
To describe the impact of persistent GERD symptoms on work productivity | Once, at first visit

CONTACTS AND LOCATIONS:
Locations (32):
- Croatia (32):
  - Research Site, Bjelovar
  - Research Site, Bulinec
  - Research Site, Crikvenica
  - Research Site, Daruvar
  - Research Site, Delnice
  - Research Site, Garešnica
  - Research Site, Gospić
  - Research Site, Ivanec
  - Research Site, Kalnik
  - Research Site, Karlovac
  - Research Site, Konjšćina
  - Research Site, Koprivnica
  - Research Site, Krapina
  - Research Site, Lovran
  - Research Site, Ludbreg
  - Research Site, Nedelišće
  - Research Site, Opatija
  - Research Site, OriovacGornja Vrba
  - Research Site, OtokPrivlakaIlokVukovarRetkovciGunjGarcin
  - Research Site, Pregrada
  - Research Site, PulaPorecPazinLabinRovinj
  - Research Site, Rijeka
  - Research Site, Samobor
  - Research Site, SenjVodiceTrogirSinjImotskiMokosicaPloceMetkovic
  - Research Site, Sisak
  - Research Site, SlavonskibrodOsijekVisnjevacKoskaDonji miholjacPleternicaVelik
  - Research Site, VarazdinCakovec
  - Research Site, Virje
  - Research Site, Zabok
  - Research Site, ZadarSibenikDubrovnik
  - Research Site, Zagreb
  - Research Site, Zlatar